CLINICAL TRIAL: NCT01373359
Title: A One Year Double Blind Randomized Controlled Trial of Sublingual Misoprostol (400 µg) Versus Intramuscular Oxytocin (10 IU) in the Prevention of Postpartum Bloodloss at KLE Hospital, Belgaum
Brief Title: Prevention of Postpartum Haemorrhage With Sublingual Misoprostol or Oxytocin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jawaharlal Nehru Medical College (Other)
Collaborators: Cipla Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Dr. M. B. Bellad, Professor, Department. of Obstetetrics. & Gynaecology, KLE University Jawaharlal Nehru Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MDC/DOME/3707
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2008-01

CONDITIONS: Postpartum Hemorrhage
Keywords: Misoprostol, oxytocin, postpartum blood loss, hemoglobin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sublingual misoprostol (Experimental): 400 µg powdered misoprostol administered sublingually; IM placebo
  Interventions: Drug: Misoprostol
- Oxytocin (Active Comparator): 10 IU IM oxytocin; placebo powder
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — 400 µg sublingual misoprostol
  Arms: Sublingual misoprostol
Drug: Oxytocin — 10 IU IM
  Arms: Oxytocin

SUMMARY:
Sublingual misoprostol produces rapid peak concentration and is more effective than oral misoprostol for prevention of excessive postpartum bleeding. The study hypothesis was to test whether women receiving sublingual misoprostol for prevention of postpartum hemorrhage have 30 ml less average blood loss than women receiving oxytocin, the standard of care for prevention of postpartum hemorrhage. We conducted a Double blind randomized controlled trial of .652 consenting, eligible pregnant women admitted to the labor room of the teaching hospital at J N Medical College, Belgaum, India. Women participating in the study were assigned by computer generated randomization to receive the study medications and placebos within one minute after clamping and cutting the umbilical cord. We also looked at the drugs effects on postpartum blood loss at or above ≥500 ml (considered hemorrhage), and the percent of women experiencing more than a 10% decline in haemoglobin, and reported drug side effects.

ELIGIBILITY:
Inclusion Criteria:

* Women with a gestational age >28weeks
* singleton pregnancy with cephalic presentation anticipating a normal spontaneous vaginal delivery (including episiotomy)
* a haemoglobin ≥ 8g/dl upon presentation who were admitted to labour room in the KLE teaching hospital attached to J N Medical College, Belgaum

Exclusion Criteria:

* Women with pregnancy induced hypertension
* antepartum haemorrhage
* previous caesarean section or presence of uterine scar
* diagnosed chorioamnionitis
* oxytocin induction or augmentation of labour
* intrauterine death
* diagnosed medical disorders (such as diabetes, cardiac, renal and hepatic diseases, etc.) or those in active labour (defined as >4 cm dilatation)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 652 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
mean blood loss | 2 hours after delivery
  Blood loss was objectively measured using the BRASSS-V DrapeTM, placed under the buttock before the delivery. The calibrated blood collection receptacle was opened after the delivery and drainage of amniotic fluid. Blood collected in the drape was transferred to measuring jar with 10 ml calibrations for accuracy. Blood soaked swabs were weighed in grams, and the known dry weight of the swabs was subtracted; this volume was added to the drape's measured blood volume (assuming 1 gm equivalence with 1 ml).
postpartum hemorrhage (Blood loss >500 mls) | 2 hours after delivery
  Blood loss was objectively measured using the BRASSS-V DrapeTM, placed under the buttock before the delivery. The calibrated blood collection receptacle was opened after the delivery and drainage of amniotic fluid. Blood collected in the drape was transferred to measuring jar with 10 ml calibrations for accuracy. Blood soaked swabs were weighed in grams, and the known dry weight of the swabs was subtracted; this volume was added to the drape's measured blood volume (assuming 1 gm equivalence with 1 ml).

SECONDARY OUTCOMES:
The percent of women experiencing a ≥10% postpartum decline in haemoglobin | At presentation for delivery and 12-48 hours after delivery
  Hemoglobin was obtained at presentation for delivery and again between 12 and 48 hours after delivery.
Medication side effects | 2 hours after delivery
  Self reported side effects including nausea, vomiting, diarrhoea, abdominal pain, shivering and elevated temperature

CONTACTS AND LOCATIONS:
Overall Officials: M B Bellad, M.D., Principal Investigator — Jawaharlal Nehru Medical College
Locations (1):
- Jawaharlal Nehru Medical College, Belagavi, Karnataka, India